CLINICAL TRIAL: NCT02163434
Title: Comparison of Gabapentin and Metoclopramide for Treating Hyperemesis Gravidarum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Thomas Guttuso, Associate Professor of Neurology, Obstetrics & Gynecology, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 496486-3; 1R01HD076313-01A1 (NIH)
Record Dates: First submitted 2014-06-09; First posted 2014-06-13 (Estimated); Results first posted 2021-09-27 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Hyperemesis Gravidarum
Keywords: pregnancy; nausea; vomiting; hyperemesis; treatment; gabapentin; metoclopramide; safety
MeSH Terms: conditions — Hyperemesis Gravidarum; Nausea; Vomiting | interventions — Gabapentin; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gabapentin (Experimental): 1800-2400mg/day divided tid or qid, orally.
  Interventions: Drug: Gabapentin
- metoclopramide (Experimental): 45-60mg/day divided tid or qid, orally
  Interventions: Drug: Metoclopramide

INTERVENTIONS:
Drug: Gabapentin
  Other Names: Neurontin
  Arms: gabapentin
Drug: Metoclopramide
  Other Names: Reglan
  Arms: metoclopramide

SUMMARY:
The investigators will compare the effectiveness of gabapentin to metoclopramide for 1 week among 60 women with hyperemesis gravidarum (HG) in this randomized, double-blinded trial. After completion of the 1-week double-blind phase, subjects will be offered open-label gabapentin with rescue metoclopramide until their symptoms no longer require treatment. Enrollment will occur at the University's at Buffalo, of Rochester and of Wisconsin.

ELIGIBILITY:
Inclusion Criteria:

1. Have received at least 2 administrations of intravenous (iv) hydration separated by at least 1 week or daily emesis for at least the last 14 days and 1 administration of iv hydration.
2. Have at least one of the following: 2-4+ ketonuria, serum potassium < 3.4mmol, or >5% weight loss from weight upon entry to prenatal care.
3. Have failed therapy with at least one antiemetic.
4. Have fetal ultrasound within 6 weeks prior to enrollment confirming a normal-appearing, intrauterine, singleton pregnancy of gestational age < 16 weeks at time of enrollment.
5. Felt by the patient's obstetrician or emergency room attending physician not to have other medical problems such as bowel obstruction, pancreatitis, biliary colic, or peptic ulcer disease that could be contributing to the patient's symptoms.
6. Be >18 years old and not decided to terminate the pregnancy.
7. Have not received or planning to receive a peripherally inserted central catheter (PIC line).
8. Have a Motherisk-PUQE score of ≥12 for the 24-hour Baseline period.
9. Felt not to have any other significant medical, psychiatric or substance abuse problem that would preclude participation in the study.
10. Denies drinking any alcohol after learning about current pregnancy.
11. Agrees to discontinue any current anti-emetic treatments (including antihistamines, ginger, > 10mg/day vitamin B6, serotonin or dopamine antagonists, anticholinergics, acupuncture, hypnosis, or wrist bands) for the next 4 weeks.
12. Pregnancy not conceived through in-vitro fertilization.
13. Able to understand and comply with the study procedures and give informed consent.

Exclusion Criteria:

None not mentioned under Inclusion Criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-06; Primary Completion 2019-10 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University at Buffalo, Buffalo, New York
  - University of Rochester, Rochester, New York

REFERENCES:
- [Background] Guttuso T Jr, Robinson LK, Amankwah KS. Gabapentin use in hyperemesis gravidarum: a pilot study. Early Hum Dev. 2010 Jan;86(1):65-6. doi: 10.1016/j.earlhumdev.2009.11.003. Epub 2009 Dec 16. PMID 20015600
- [Background] Holmes LB, Hernandez-Diaz S. Newer anticonvulsants: lamotrigine, topiramate and gabapentin. Birth Defects Res A Clin Mol Teratol. 2012 Aug;94(8):599-606. doi: 10.1002/bdra.23028. Epub 2012 Jun 22. PMID 22730257
- [Background] Guttuso T Jr. Gabapentin's anti-nausea and anti-emetic effects: a review. Exp Brain Res. 2014 Aug;232(8):2535-9. doi: 10.1007/s00221-014-3905-1. Epub 2014 Mar 26. PMID 24668130
- [Derived] Guttuso T Jr, Messing S, Tu X, Mullin P, Shepherd R, Strittmatter C, Saha S, Thornburg LL. Effect of gabapentin on hyperemesis gravidarum: a double-blind, randomized controlled trial. Am J Obstet Gynecol MFM. 2021 Jan;3(1):100273. doi: 10.1016/j.ajogmf.2020.100273. Epub 2020 Oct 29. PMID 33451591

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin: 1800-2400mg/day divided tid or qid, orally.
  Gabapentin
- Metoclopramide: 45-60mg/day divided tid or qid, orally
  Metoclopramide
Period: Overall Study
Arm/Group | Gabapentin | Metoclopramide
Started | 15 | 16
Completed | 12 | 9
Not Completed | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Metoclopramide | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (5.9) | 26.3 (3.9) | 26.25 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  non-Hispanic white | 2 | 2 | 4
  non-Hispanic black | 10 | 6 | 16
  Hispanic white | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Baseline Adjusted Mean Daily Motherisk-PUQE Total Scores (Pregnancy-unique Quantification of Emesis and Nausea Scale) for Days 5-7
Description: Score range: 6-30 with higher score indicating a worse outcome.
Time Frame: 1 week
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Gabapentin | Metoclopramide
Number analyzed (Participants) | 12 | 9
units on a scale | 6.35 (2.44) | 13.22 (2.39)
Statistical Analysis 1: Comparison: Gabapentin vs Metoclopramide; Test type: Superiority; p = 0.01, Mixed Models Analysis

2. Secondary Outcome: Baseline Adjusted Mean Daily Nausea Scores From the Motherisk-PUQE for Days 5-7.
Description: Score range: 2-10 with higher score indicating a worse outcome.
Time Frame: 1 week
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Gabapentin | Metoclopramide
Number analyzed (Participants) | 12 | 9
units on a scale | 2.01 (0.45) | 3.69 (0.45)
Statistical Analysis 1: Comparison: Gabapentin vs Metoclopramide; Test type: Superiority; p = 0.005, Mixed Models Analysis

3. Secondary Outcome: Baseline Adjusted Mean Daily Oral Nutrition Score for Days 5-7
Description: Score range: 0-15 with higher score indicating a better outcome.
Time Frame: 1 week
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Gabapentin | Metoclopramide
Number analyzed (Participants) | 12 | 9
units on a scale | 7.86 (1.23) | 4.01 (1.34)
Statistical Analysis 1: Comparison: Gabapentin vs Metoclopramide; Test type: Superiority; p = 0.01, Mixed Models Analysis

4. Secondary Outcome: Percent of Subjects Requiring Repeat iv Hydration or Hospital Admission for HG From the Outpatient Setting.
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Metoclopramide
Number analyzed (Participants) | 12 | 9
Participants | 5 | 5

5. Secondary Outcome: Global Satisfaction of Treatment at the Study Endpoint.
Description: Score range: 0-4 with higher score indicating a better outcome.
Time Frame: 1 week
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Gabapentin | Metoclopramide
Number analyzed (Participants) | 12 | 9
units on a scale | 2.22 (1.56) | 0.63 (0.74)
Statistical Analysis 1: Comparison: Gabapentin vs Metoclopramide; Test type: Superiority; p = 0.03, Mixed Models Analysis

6. Secondary Outcome: Desire to Continue Therapy at Study Endpoint
Description: Scores: 0=no, 1=yes. Thus, a higher score indicates a better outcome.
Time Frame: 1 week
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Gabapentin | Metoclopramide
Number analyzed (Participants) | 12 | 9
units on a scale | 0.67 (0.50) | 0.14 (0.38)
Statistical Analysis 1: Comparison: Gabapentin vs Metoclopramide; Test type: Superiority; p = 0.06, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 1 week of double-blind therapy
Arm/Group | Gabapentin | Metoclopramide
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 4/15 | 3/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=15) | Metoclopramide (N=16)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hot Flashes (Endocrine disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT02163434/Prot_SAP_000.pdf